CLINICAL TRIAL: NCT03807687
Title: Registry of Subjects Affected by Pancreatic Disease and Evaluated at the Pancreas Institute of Verona
Brief Title: Registry of Pancreatic Disease
Acronym: PAD-R
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: PAD-R 1101CESC
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Diseases; Pancreatic Neoplasms; Pancreatitis
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Neoplasms; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 27 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with pancreatic disease: Patients diagnosed with pancreatic disease evaluated at this institution.

SUMMARY:
This clinical data registry records information about the health status and healthcare performances received by participants affected by every type of pancreatic disease or disorder. All data (demographic, clinical, biochemical, radiological, pharmacological, genetic...) and audio and/or video recording from operative room are collected in order to be used for prospective or retrospective studies.

ELIGIBILITY:
Inclusion Criteria:

* any type of pancreatic disease: inflammatory and neoplastic (including solid and cystic lesions)

Exclusion Criteria:

* physically or mentally inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient affected by pancreatic disease admitted to General and Pancreatic Surgery Department of Verona University Hospital from 01/01/1990 to 12/01/2046
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2046-12-01 (Estimated); Study Completion 2046-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Survival from Diagnosis to time of death

SECONDARY OUTCOMES:
Postoperative morbidity | 90 days
  Occurrence of Pancreatic Fistula, Biliary fistula, Enteric fistula, Delayed Gastric Emptying, Hemorrhage or Sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassi, Prof, Principal Investigator — AOUI Verona
Locations (1):
- AOUI Verona, Verona, Italy